CLINICAL TRIAL: NCT05183048
Title: Comparison of 89Zr Panitumumab and (18)F-Fluorodeoxyglucose to Identify Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Suzanne E. Lapi, PhD, Professor, Advanced Imaging Facility, Division of Advanced Medical Imaging Research, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300008612; UAB Radiology Pilot Grant (Other: UAB Radiology)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [89Zr]panitumumab-PET/MRI patients (Experimental): All study patients will receive [89Zr]Panitumumab-PET/MRI imaging.
  Interventions: Drug: [89Zr]Panitumumab Tracer

INTERVENTIONS:
Drug: [89Zr]Panitumumab Tracer — All patients entered into the study will have [89Zr]Panitumumab-PET/MRI imaging.

SUMMARY:
This pilot clinical study will investigate if Zirconium-89 (89Zr) panitumumab- Positron Emission Tomography/ Magnetic Resonance Imaging (PET/MRI) imaging can more accurately determine size and location of primary tumors compared to standard of care Fludeoxyglucose (18F-FDG) -PET/MRI in newly diagnosed patients with head and neck squamous cell carcinoma (HNSCC) who are undergoing surgical resection. This study is for imaging purposes only and is not a treatment study. The results of this study will not change the clinical treatment plan.

DETAILED DESCRIPTION:
The study is an open label, single center, non-randomized, pilot study to determine the efficacy of [89Zr]panitumumab to localize primary tumor in patients with squamous cell carcinoma of the head and neck (HNSCC) that undergo surgery with curative intent compared to standard of care,18F-FDG. Enrolled subjects are clinically and radiographically node negative (cN0) based on the preoperative work-up, which includes a standard of care physical exam and evaluation of the pre-existing imaging data (CT or MRI scan, which may be collected before or during standard of care [18F]FDG imaging).

Consenting and Screening phone call

Physicians who are study sub-investigators will identify and discuss the study with eligible patients they see in clinic. If interested in the study, sub-investigators will contact study coordinators to discuss further with patients. Interested participants will be consented prior to any study procedures. Consent may be signed during clinical visit or at a more convenient time by the participant.

Enrolled patients will be called to discuss the study and complete an MRI screening form. Participants meeting MRI screening criteria will be scheduled for the first visit.

Visit 1 (within 5-9 days prior to surgery)

During the first visit, consented participants will have a standard of care FDG-PET/MRI, if not already performed, vital signs checked, a 50 mg infusion of panitumumab, and a 1.5 millicurie(mCi) injection of [89Zr]panitumumab. No special patient preparation is required.

FDG-PET/MRI administration and imaging:

[18F]FDG is an FDA approved radiopharmaceutical and is used as per standard of care in this study. [18F]FDG will be obtained from a commercially licensed Radiopharmacy for this study.

If the PET/MRI is unavailable or contraindicated for a participant, FDG-PET/CT may be used at the discretion of the investigator and study radiologist.

Panitumumab administration:

Participants will receive an intravenous infusion of 50 mg dose of panitumumab over 10 minutes to minimize uptake of the radiotracer in normal tissues. The administration of a fixed small dose of unlabeled antibody to improve tumor-to-normal-tissue (T/N) uptake of the radiolabeled antibody is standard in this type of imaging procedure. Infusion of panitumumab will be prepared by the research pharmacy and administered in the Clinical Research Unit (CRU) infusion area of the Jefferson Tower (JT) according to normal treatment protocol by Oncology personnel appropriately trained and certified to administer chemotherapeutic agents. Following the infusion of panitumumab, participants will be monitored for approximately 30 minutes for infusion reactions and side effects.

Because the dose of panitumumab being administered is a fraction, about 1/7 of the dose normally administered as standard treatment, and it is being administered one time per study, no dose modifications for panitumumab are allowed. We do not expect any side effects as a result of the administration of the small dose of panitumumab for this study. However, as it is suggested for therapeutic dose, participants who experience severe dermatological toxicity (National Cancer Institute Common Terminology Criteria (NCI-CTC) grade 3 and higher) or serious infusion reaction (i.e., dyspnea, chest tightness, fever, rigors or hypotension) during panitumumab administration will have the infusion stopped and will be excluded from further participation in the study. Continuation of dosing and continuation in study will be based on the severity and resolution of the event and will be at the discretion of the investigator and the referring/treating physician. Any treatment for an infusion reaction will be administered per institutional practices.

[89Zr]Panitumumab administration: At least 60 minutes after injection of panitumumab, participants will receive an injection of [89Zr]Panitumumab in the Advanced Imaging Facility. The administered dose will be 1.5 mCi (±10%) at the time of injection. The amount of injected drug is <1 mg of Panitumumab. The administered intravenous volume of [89Zr]Panitumumab is ≤ 10 mL and will be infused over approximately 1 minute, followed by a saline flush. The infusion will be terminated in any patient who exhibits anaphylaxis, significant dyspnea, or chest pain. Participants will be monitored for 30 minutes after injection.

The adverse events to be specifically monitored during the infusions include localized discomfort at the IV injection sites, pain, respiratory difficulties, flushing, dizziness, pruritus/rash, and any other symptoms that could be secondary to an anaphylactic reaction. The subject will be instructed to report any subjective symptoms or sensory changes noted. Participants will be called by study staff within 48 hours to ask about any signs of adverse effects.

Visit 2 (within 3-5 days prior to surgery and 2-4 days after [89Zr]Panitumumab injection)

Participants will return to the The University of Alabama at Birmingham (UAB) Advanced Imaging Facility for [89Zr]panitumumab-PET/MRI imaging 2 to 4 days after receiving the radiopharmaceutical. Imaging will include a scan of the head and neck region (static) continuing with vertex-to-thigh. No special patient preparation will be requested (i.e., fasting or hydration) on the day of the scans. All participants will be scanned with a calibrated PET/MRI scanner (GE SIGNA 3.0 Tesla PET/MRI scanner; GE Healthcare, Chicago, IL) in the three-dimensional mode. The PET images will be processed using a dedicated workstation (MIM software; MIM, Cleveland, Ohio or Advantage Workstation; GE Healthcare, Chicago, IL). Images will be analyzed by a nuclear medicine physician who will be blinded from the clinical information on target lesion distribution. Investigator (CoI: Dr. McConathy) blinded to the imaging agent used (FDG or [89Zr]panitumumab) and to clinical disease status will visually inspect de-identified PET/MRI images and draw regions of interest (ROI's) over suspicious lesions. Image processing software will calculate standard uptake value (SUV)max and Tumor to background radio (TBR) values.

If the PET/MRI is unavailable or contraindicated for a participant, the PET/CT may be used at the discretion of the investigator and study radiologist.

Standard of Care Surgical Resection and Follow up

Patients will undergo standard of care surgical resection as directed by treating physician. Histological assessments and other post-surgical information will be obtained by follow up review of patient's medical records.

Histological assessment Routine H&E staining will be performed for histological assessment by a board-certified pathologist to determine the presence/absence of tumor and tumor dimensions. Findings will be compared to PET imaging findings. Subsequently, histological findings will be correlated with autoradiography findings using slide-mounted sections obtained from paraffin-embedded blocks. Immunohistochemistry on unstained lymph node sections will be performed to evaluate Estimated Glomerular Filtration Rate (eGFR) expression, tumor density (anti-pan cytokeratin), vessel density, and histiocyte presence. For the latter we will look amongst others at macrophages, T- and B-cells. Stained slides will be imaged using the Bio-Imagene (Ventana Medical Systems) optical scanner. Findings will then be correlated to the PET imaging results. Additional sections will be collected as needed.

Clinical and pathological response data will be collected at the end of the treatment period. Once the data is collected, no further follow up will be required for the patients.

Future Use of Stored Specimens and Data

Data and samples collected for this study will be analyzed and stored on site. After the study is completed, the de-identified, archived data will be stored on site, for use by other researchers including those outside of the study if participant allows. With participant approval, when the study is completed, access to study data and/or samples will be provided through the Volker Hall Tissue Bank.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed diagnosis of squamous cell carcinoma of the head and neck
2. Subjects newly diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection.
3. Subjects are to be staged clinically and radiographically node negative (cN0)
4. Planned standard of care surgery with curative intent for squamous cell carcinoma
5. Age > 18 years
6. Have acceptable hematologic status, coagulation status (11 to 13.5 seconds. international normalized ratio (INR) of 0.8 to 1.1), kidney function, and liver function including the following clinical results:

   1. Hemoglobin ≥ 9 gm/dL
   2. White blood cell count ≥ 3000/mm3
   3. Platelet count ≥ 100,000/mm3
   4. Serum creatinine ≤ 1.5 times upper reference range
   5. alanine transaminase (ALT) (SGPT) 7-56 units/liter, aspartate aminotransferase (AST) (SGOT) 5-40 units/liter.

Exclusion Criteria:

1. Received an investigational drug within 30 days prior to the first dose of [89Zr]panitumumab.
2. Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment.
3. Previous HNSCC resection.
4. History of infusion reactions to monoclonal antibody therapies.
5. Pregnant or breast-feeding women.
6. Magnesium (<1.7 mg/dL) or potassium (<3.6 mmol/L) lower than the normal institutional values.
7. Subjects receiving Class I-A (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
8. Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
9. Severe renal disease or anuria (Creatinine within normal institutional limits OR Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels).
10. Known hypersensitivity to panitumumab or any of its components.
11. Weight over 350 lbs., due to the scanner bore size.
12. Contraindication for MRI procedures (e.g. non-removable metal implants or certain tattoos).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Image Quality | 5-9 days prior to surgery
  Diagnostic image quality of [89Zr]Panitumumab PET imaging in patients with newly diagnosed HNSCC. Standardized Uptake Values (SUVs) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lapi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No